CLINICAL TRIAL: NCT03582332
Title: Effect of Continuous Administration of Different Therapeutic Dosages of Indomethacin and Etoricoxib in the Management of Axial Spondyloarthritis: A Randomized Controlled Trial
Brief Title: Serum Creatinine Change / Renal Adverse Effect With Use of Non-steroidal Painkillers in Axial Spondyloarthritis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Khandker Mahbub-Uz-Zaman, Resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2015/5965
Record Dates: First submitted 2018-03-12; First posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — Capsules; Indomethacin; Etoricoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A in phase 1 (Active Comparator): Indomethacin 75 mg, extended release capsule twice daily
  Interventions: Drug: Indomethacin SR, 75 Mg Oral Capsule, Extended Release
- Group B in phase 1 (Active Comparator): Indomethacin 25 mg capsule, 2 capsule twice daily
  Interventions: Drug: Indomethacin 25 Mg Oral Capsule
- Group A in phase 2 (Active Comparator): Etoricoxib 90 mg once daily
  Interventions: Drug: Etoricoxib 90 mg
- Group B in phase 2 (Active Comparator): Etoricoxib 60 mg once daily
  Interventions: Drug: Etoricoxib 60 mg

INTERVENTIONS:
Drug: Indomethacin SR, 75 Mg Oral Capsule, Extended Release — Indomethacin SR, 75 Mg Oral Capsule, Extended Release orally twice daily
  Other Names: indomethacin
  Arms: Group A in phase 1
Drug: Indomethacin 25 Mg Oral Capsule — Indomethacin 25 Mg Oral Capsule, 2 capsule orally twice daily
  Other Names: indomethacin
  Arms: Group B in phase 1
Drug: Etoricoxib 90 mg — Etoricoxib 90 mg once daily orally
  Other Names: Etoricoxib
  Arms: Group A in phase 2
Drug: Etoricoxib 60 mg — Etoricoxib 60 mg once daily orally
  Other Names: Etoricoxib
  Arms: Group B in phase 2

SUMMARY:
2 Non-steroidal anti-inflammatory drugs (NSAIDs), indomethacin and etoricoxib were prescribed sequentially in Axial Spondyloarthritis patients according to the internationally accepted guidelines to determine serum creatinine change with NSAIDs use.

DETAILED DESCRIPTION:
The study had 2 phases. In phase 1, Patients of axial Spondyloarthritis were randomized into 2 groups; group A and group B. they were put on indomethacin 150 mg/day and indomethacin 100 mg/day respectively and were followed up at 3rd week. Those who had normal serum creatinine and responded with the drug were followed up to 24th week. Those who did not respond were excluded from phase 1 and were enrolled in phase 2. Non-responders of indomethacin 150mg and indomethacin 100 mg were put on etoricoxib 90 mg and etoricoxib 60 mg respectively. Again followed up to 24th week.

ELIGIBILITY:
Inclusion Criteria:

* SpA (axial) patients according to Assessment of Spondyloarthritis International Society (ASAS) criteria with BASDAI > 4

Exclusion Criteria:

* Inadequate response to therapeutic dose of indomethacin or etoricoxib, taken for at least 2 weeks continuously
* Abnormal serum creatinine : serum creatinine >1.3 mg/dl
* Abnormal SGPT: SGPT > 40 U/L
* Hypertension: Systolic blood pressure > 140 mm Hg and/ or diastolic blood pressure >90 mm Hg or on anti-hypertensive drug
* Dyspepsia or active peptic ulcer disease : upper abdominal discomfort or upper abdominal pain related with food or peptic ulcer disease diagnosed by upper gastrointestinal endoscopy
* Diabetes mellitus: abnormal random plasma glucose or diagnosed case of diabetes mellitus
* Ischemic heart disease: history of angina or ECG changes suggestive of ischemic heart disease
* Active congestive heart failure: pedal edema with tender hepatomegaly with raised JVP or diastolic dysfunction on echocardiography
* Asthma: diagnosed case of asthma or rhonchi on chest auscultation
* Bleeding problems: having a history of prolonged bleeding
* Pregnancy: missed period followed by positive pregnancy test
* Simultaneous use with certain medications such as warfarin, phenytoin, cyclosporine, probenecid, lithium, digoxin, ACE inhibitor, thiazide

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2016-06-23 (Actual); Study Completion 2016-06-23 (Actual)

PRIMARY OUTCOMES:
Serum creatinine change | 3rd week and 24th week
  change in serum creatinine >25% from baseline with use of indomethacin and etoricoxib in Axial Spondyloarthritis patients

SECONDARY OUTCOMES:
Bath Ankyiosing Spodylitis Disease Activity Index (BASDAI) | 3rd week and 24th week
  <4 responded to treatment, 4 or more means not responded to treatment
Ankylosing Spondylitis Disease Activity Score (ASDAS) | 3rd week and 24th week
  ASDAS: <1.3 between "inactive disease" and "moderate disease activity", <2.1 between "moderate disease activity" and "high disease activity", and >3.5 between "high disease activity" and "very high disease activity"

CONTACTS AND LOCATIONS:
Overall Officials: Khandker Mahbub-Uz-Zaman, MD, Principal Investigator — Resident

IPD SHARING:
Plan to Share IPD: Undecided